CLINICAL TRIAL: NCT00409747
Title: Treatment of Childhood Regressive Autism With Minocycline: an Anti-Inflammatory Agent Active Within the CNS
Brief Title: Minocycline to Treat Childhood Regressive Autism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070024; 07-M-0024 (Other: NIH Protocol number)
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Autism; Minocycline; Regressive Autism
Keywords: Immunology; Microglia; NF-Kappa-B; Antibiotic; Autism; Minocycline; Regressive Autism
MeSH Terms: conditions — Autistic Disorder; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline (Experimental)
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline

SUMMARY:
There is a subgroup of children with autism that appears to develop typically for a period of time, and then loses social or language skills, or regresses. A recent study by Vargas and co-workers at Johns Hopkins has demonstrated that this regressive type of autism is associated with chronic brain inflammation as shown by an abnormal production of inflammatory cytokines among other abnormalities.

This present study will test the effectiveness of minocycline, an antibiotic with anti-inflammatory properties, in treating regressive autism. Although behavioral therapies have improved some symptoms of autism, there are no medical treatments for the disorder, and many children have ongoing behavioral difficulties. A medicine with anti-inflammatory properties may be beneficial for children with regressive autism.

This will be an open-label trial, meaning all children in this study will receive minocycline. They will also receive vitamin B6 to reduce the possible chance of side effects of the minocycline.

Children ages 3 to 12 with regressive autism may be eligible for this study. The children will take minocycline and vitamin B6 daily for 6 months. Prior to starting the medication and vitamin B6, children will receive a comprehensive diagnostic assessment for autism as well as a physical examination, medical history, and laboratory tests. Children will then receive ongoing assessments to monitor their behavior, communication, language skills, and medical issues at 2 weeks, and at 1, 2, 4, 6, and 12 months. Children who respond to the treatment will receive an additional 3 months of minocycline and vitamin B6.

DETAILED DESCRIPTION:
Autism is a neurodevelopmental disorder that results in abnormalities of social and language development and is associated with rigid and repetitive behaviors. Although there is strong evidence of heritability, the involved genes have not been identified. The prevalence of autism spectrum disorders may be as common as 1 in 166. The average concordance rate in monozygotic twins is 70% suggesting that environmental factors play a role in the disease. Subgroups of autistic children seem unusually sensitive to infections, immunizations and dietary factors, but none of these factors has been causally identified with the disease. Nevertheless, autoimmunity has been considered to play a role on the basis of indirect evidence. There is no evidence-based efficacious treatment for autism.

There is a subgroup of children with autism that appear to develop typically for a period of time, and then lose skills, or regress. A recent study by Vargas and co-workers at Johns Hopkins has demonstrated that the regressive subtype of autism is associated with chronic brain neuroinflammation as exemplified by activation of microglia and astroglia and the abnormal production of inflammatory cytokines and growth factors assayed in both tissue samples (brain banks) and CS. The authors remarked that these responses were similar to those seen in some neurodegenerative disorders such as amyotrophic lateral sclerosis, and that chronic microglia activation appears to be responsible for a sustained neuroinflammatory response that facilitates the production of multiple neurotoxic mediators. Chronic neuroglial activation could be the result of an abnormal persistence of a fetal development pattern. In this scenario neuroglial activation could play a role in initiating and in maintaining the pathology. Alternatively, neuroglial activation may only be a secondary response to the initiating causal factor(s) and not a direct effector of injury. Since neuroglial activation requires the nuclear translocation of the pro-inflammatory transcription factor NF-kappa B, and since inhibitors of NF-kappa-B with good CNS penetrance are available, the role of neuroinflammation in initiating and sustaining the autistic condition can be probed.

The antibiotic minocycline is a powerful inhibitor of microglial activation, apparently through blockade of NF-kappa-B nuclear translocation. Minocycline is neuroprotective in mouse models of amyotrophic lateral sclerosis (ALS) and Huntington's disease and has been recently shown to stabilize the course of Huntington's disease in humans over a 2-year period.

To evaluate the possibility of benefit in autistic children, we propose to conduct an open-label trial of the anti-inflammatory antibiotic minocycline, an agent that reduces inflammation by blocking the nuclear translocation of the proinflammatory transcription factor NF-kappa-B. Minocycline is Food and Drug Administration (FDA)-approved for treatment of a variety of infections and has been widely used for the treatment of adolescent acne. Minocycline is currently in phase III trials for the treatment of Huntington's disease and amyotrophic lateral sclerosis.

This proposal is for an initial 6-month, single-arm, off label, open-label study (with a 3 month extension phase offered to responders) that will evaluate dose safety and efficacy of minocycline in 10 children, ages 3 to 12 years, with a primary diagnosis of autism and a history of developmental regression. The subjects will be evaluated by a diagnostic/behavioral assessment, and the extent of neuroinflammation judged by CSF cytokine/chemokine profiles before and after the 6-month treatment. Subjects will also be given 0.6 mg/kg vitamin B6 twice a day as a prophylactic for possible minocycline induced nausea and vomiting. If the results of this feasibility study are encouraging, we expect to conduct a double-blind, placebo-controlled trial of minocycline therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

The sample will be children with:

* Diagnosis of idiopathic autism and regression
* Age between 3 and 12 years
* Willingness to undergo lumbar puncture for evaluation of proinflammatory CSF cytokines
* Stable behavioral plus or minus medication therapies.

EXCLUSION CRITERIA:

* Significant prematurity at birth (less than 32 weeks gestation); or birthweight significantly below normal for gestational age (SGA--small for gestational age).
* Neurologic disorders including cerebral palsy, uncontrolled epilepsy, and Landau-Kleffner syndrome.
* Evidence of renal insufficiency or hepatic disease (to reduce the incidence of side-effects, since minocycline is excreted by the kidneys following hepatic metabolism)
* Increased risk of developing lupus-like syndrome with minocycline administration (positive anti-double stranded DNA or anti-nucleosome antibody tests at baseline, or presence of a first degree relative with S.L.E.)
* Recent (less than two months prior to study entry) initiation of a behavioral therapy program or new psychotropic medication trial.
* Subjects on one of the medications/supplements listed as those with possible interactions or those on high dose B6 supplementation. For those families who are interested in the study but are on any of these medications/supplements at the time of intake, they will be instructed to wean the medication as appropriate (working with the prescribing MD), and they will be enrolled after a 6-week wash-out period.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2006-11; Primary Completion 2010-06 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Auld DS, Robitaille R. Glial cells and neurotransmission: an inclusive view of synaptic function. Neuron. 2003 Oct 9;40(2):389-400. doi: 10.1016/s0896-6273(03)00607-x. PMID 14556716
- [Background] Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. Am J Ment Defic. 1985 Mar;89(5):485-91. PMID 3993694
- [Background] Barger SW, Moerman AM, Mao X. Molecular mechanisms of cytokine-induced neuroprotection: NFkappaB and neuroplasticity. Curr Pharm Des. 2005;11(8):985-98. doi: 10.2174/1381612053381594. PMID 15777249
- [Derived] Lane R, Kessler R, Buckley AW, Rodriguez A, Farmer C, Thurm A, Swedo S, Felt B. Evaluation of Periodic Limb Movements in Sleep and Iron Status in Children With Autism. Pediatr Neurol. 2015 Oct;53(4):343-9. doi: 10.1016/j.pediatrneurol.2015.06.014. Epub 2015 Jun 26. PMID 26231264
- [Derived] Pardo CA, Buckley A, Thurm A, Lee LC, Azhagiri A, Neville DM, Swedo SE. A pilot open-label trial of minocycline in patients with autism and regressive features. J Neurodev Disord. 2013;5(1):9. doi: 10.1186/1866-1955-5-9. Epub 2013 Apr 8. PMID 23566357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Referrals accepted from community physicians and self(parent) referrals.
Pre-assignment Details: Three subjects did not start the drug due to abnormal MRI,initial elevated liver enzymes, and and initial elevated amylase. 11 subjects began taking drug. One subject withdrew after starting drug.
Groups:
- Minocycline: Open-label minocycline treatment at 1.4 mg/kg/day
Period: Overall Study
Arm/Group | Minocycline
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 10 subjects completed the trial and had analyzable data at the 6 month mark. One child had csf collected after 3 months.
Arm/Group | Minocycline
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.2 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: z Score
Description: The Mann-Whitney U-test was used to compare pre-/post-treatment differences in analyte concentrations in serum, plasma and CSF. The Mann-Whitney U test generates a z-score test statistic with an associated p value. A negative z-statistic reflects a decrease in analyte level from pre- to post-treatment. Statistical significance level was set at 0.05. There is one test statistic (z-score) per analyte, reflecting the pre-post comparison across all subjects.
  Pre and post treatment measurements of csf analytes: TNF alpha, Il-6, CCL-2(MCP-1), CCL3 (MIP-1alpha), CCL5(RANTES), CXCL(IL-8), BDNF, CD40L, GDNF, HGF, Leptin
Time Frame: Pre and post treatment with minocyline at 6 months for 10 subjects
Population: 10 subjects completed six months of minocycline and have pre-/post-minocycline CSF samples for analysis.
Measure: Number; unit: Z-score
Arm/Group | Minocycline
Number analyzed (Participants) | 10
Z-score
  TNFalpha | -0.45
  IL-6 | -0.36
  CCL2(MCP-1) | -1.78
  CCL3(MIP-1alpha) | -0.18
  CCL5(Rantes) | -0.73
  CXCL8(IL-8) | -0.45
  BDNF | -2.03
  CD40L | -0.89
  GDNF | -0.37
  HGF | -2.19
  Leptin | -1.48

2. Secondary Outcome: Clinical Global Impressions Scale-Severity (CGI). (Connors & Barkley, 1985)
Description: This instrument has two scales - Severity (CGI-S). The CGI-S is a seven point scale with a minimum score of 1 and a maximum score as 7 as follows: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients.
Time Frame: Baseline and 6 months
Population: All children completing 6 months of drug and participating in final evaluation
Measure: Mean (Standard Deviation); unit: mean scores on global impression scale
Arm/Group | Minocycline
Number analyzed (Participants) | 10
mean scores on global impression scale
  Baseline | 4.4 (0.8)
  6 months | 4.6 (.81)

ADVERSE EVENTS:
Time Frame: 6 months of minocycline administration
Arm/Group | Overall Study/Minocycline
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study/Minocycline (N=11)
Vomiting and fever (Gastrointestinal disorders) | 1 (1) — Related to intercurrent illness

LIMITATIONS AND CAVEATS:
Small, uncontrolled pilot.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes